CLINICAL TRIAL: NCT05313009
Title: A Phase Ib / II Trial of Tarloxotinib and Sotorasib in Patients With KRAS G12C Mutations
Brief Title: Tarlox and Sotorasib in Patients With KRAS G12C Mutations
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study drug was discontinued by manufacturer for business reasons.
Sponsor: Medical University of South Carolina (Other)
Collaborators: Rain Oncology Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 103408
Record Dates: First submitted 2022-02-14; First posted 2022-04-06 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sotorasib

STUDY DESIGN:
Intervention Model Description: (1) Safety lead-in: A minimum of 6 patients and as many as 18 patients will be enrolled in a safety lead-in cohort to evaluate the safety of the combination of tarloxotinib and sotorasib. (2) Dose expansion: Once the tarloxotinib RP2Dc is reached, an expansion cohort of up to 12 patients will be enrolled to evaluate the safety of the combination of tarloxotinib and sotorasib.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- STAGE 1: SAFETY LEAD IN (n=6-18, depending on number of DLs explored) (Experimental): SAFETY LEAD IN (n=6-18, depending on number of DLs explored) 3+3 design dependent on DLTs
  Interventions: Drug: Sotorasib and Tarloxotinib
- STAGE 2: EFFICACY (n=12) (Experimental): EFFICACY (n=12)
  Interventions: Drug: Sotorasib and Tarloxotinib

INTERVENTIONS:
Drug: Sotorasib and Tarloxotinib — Sotorasib 960 mg PO daily + tarloxotinib 150 mg/m2 IV weekly
Drug: Sotorasib and Tarloxotinib — Sotorasib 960 mg PO daily + tarloxotinib IV weekly at the combination RP2D (RP2Dc).

SUMMARY:
This is a Phase IB dose expansion trial with safety lead-in evaluating the safety, clinical activity/efficacy of the combination of tarloxotinib and sotorasib in patients with KRAS G12C mutation who have progressed on any small molecule targeting KRAS G12C mutant Non-Small Cell lung cancer.

DETAILED DESCRIPTION:
KRAS acts as a key protein in transducing signals from cell surface receptors, such as receptor tyrosine kinases (RTKs) into cells to initiate a network of cytoplasmic and nuclear signaling cascades that mediate key processes, such as cell cycle entry and cell survival that regulate normal tissue homeostasis. Due to the central importance of KRAS in mediating critical cellular processes, there are significant interconnected signaling feedback pathways that protect normal cells from uncontrolled proliferation and cell death. These signaling feedback pathways are also activated by tumor cells upon inhibition of mutated KRAS, which may result in intrinsic or acquired resistance to small molecule KRAS G12C inhibitors. Pre-clinical studies in non-small cell lung cancer (NSCLC) have shown that a key pathway that may be activated upon KRAS inhibition is the upstream ERBB RTKs, which provides the rationale for dual KRAS and ERBB blockade in overcoming resistance mechanisms in KRAS mutated NSCLC.

Lung cancer is the second most common cancer and the leading cause of cancer death in the United States. There were approximately 247,270 new cases of lung cancer that occurred in 2020. Prior studies have reported that lung cancer resulted in more deaths than breast cancer, prostate cancer, colorectal cancer, and leukemia combined in men ≥40 years old and women ≥60 years old. The past decade has seen a revolution of new advances in the management of non-small cell lung cancer (NSCLC) with remarkable progresses in screening, diagnosis, and treatment. The advances in systemic treatment have been driven primarily by the development of molecularly targeted therapeutics, immune-checkpoint inhibitors and anti-angiogenic agents, all of which have transformed this field with significantly improved patient outcomes. Despite these advances, most patients with advanced NSCLC have incurable disease, particularly after failure of a platinum-based chemotherapy regimen and check point inhibitors.

One of the earliest identified molecular drivers of NSCLC is the GTPase transductor protein called KRAS. It is a member of the RAS family of oncogenes and at the apex of multiple signaling pathways central to tumor cell proliferation. KRAS mutant lung cancers have worse outcomes in both early stage and advanced metastatic settings, illustrating the critical need for novel agents targeting KRAS-driven NSCLC. KRAS G12C mutations are present in ~15% of lung adenocarcinomas and 0-8% of other cancers. The missense mutation at codon 12 interferes with the GTPase, activating protein mediated GTP hydrolysis and shifting the equilibrium between the signaling-competent KRAS-GTP and signaling incompetent KRAS-GDP in favor of the GTP bound state. This process links upstream cell surface receptors such as the ERBB family (EGFR, HER-2, HER-3, HER-4) to downstream pathways such as RAF/MEK/ERK and PI3K/AKT/mTOR which leads to uncontrolled cell proliferation and survival.

Attempts to identify small molecular inhibitors of KRAS have been unsuccessful for many years as there was a lack of a clearly defined deep pocket in the structure of RAS outside of the nucleotide binding site and the challenge of targeting the nucleotide binding site due to extraordinarily high affinity of GTP. Recently, several pioneering studies have identified small molecule cysteine-reactive inhibitors that covalently modify the mutant KRAS G12C protein to reveal an allosteric switch II pocket. The induction of the structurally disordered pocket by these small molecule inhibitors converts the GTP preference of naïve KRAS G12C to the inactive GDP bound state, impairing its interaction with downstream effectors.

AMG510/Sotorasib was the first KRAS G12C inhibitor to the enter the clinic. A Phase I/II clinical trial involving 129 patients included 59 patients with KRAS G12C mutated NSCLC who had progressed on prior standard therapies. Patients were enrolled in dose escalation and expansion cohorts to receive daily sotorasib monotherapy (960 mg PO daily). At a median follow up of 12.2 months, approximately 50% of NSCLC patients demonstrated tumor regression with a confirmed objective response rate (ORR) of 37.1% (95% CI 28.6-46.2%) and a disease control rate (DCR) of 80.6% (95% CI 72.6-87.2%). The median time to objective response was 1.4 months and median duration of response was 10 months, with median progression free survival (PFS) of 6.8 months. The FDA has now accepted a new drug application and granted it a priority review for the treatment of patients with KRAS G12C mutant locally advanced or metastatic NSCLC following at least 1 prior systemic treatment, with an expected decision date by August 2021.

Although the results from these early-stage clinical trials showed promise, ~50% of KRAS G12C mutant NSCLC patients failed to respond to therapy and rate of relapse is high calling for the need for novel combinations to overcome intrinsic and acquired resistance mechanisms in this subset of patients.

It was previously thought that constitutively active oncogenic KRAS induces growth factor independence. However, recent evidence has suggested that specific KRAS mutant isoforms such as KRAS G12C may be regulated by upstream activation of several receptor tyrosine kinases. The pattern of RTK dependence appears to vary between KRAS G12C mutant cancer but numerous RTKs are involved in the adaptive feedback mechanism to G12C inhibition. This may be mediated through an adaptive RAS pathway activation. Silencing oncogenic KRAS in EGFR/HER dependent cells reduced cellular growth and induced a modest apoptotic signal. The depletion of KRAS expression by mutant specific siRNA was accompanied by a reduction in AKT phosphorylation in the ERBB dependent subset and activation of STAT3, which suggests a feedback loop via STAT3 that re-establishes oncogenic signaling thereby compensating for the loss of AKT survival signals. Pan ERBB inhibition in these KRAS G12C mutated NSCLC lines resulted in a potent suppression of growth and inhibition of receptor signaling and downstream signaling effectors. Thus, sole silencing of oncogenic KRAS may not be an effective therapeutic strategy in KRAS-addicted cancers since upstream events and feedback loops are likely to attenuate or annul the effects of the therapeutic intervention.

These pre-clinical studies provide a solid ground to evaluate the use of pan-ERBB inhibitors in combination with KRAS G12C inhibitors in patients with KRAS mutant lung tumors.

Tarloxotinib is a recently discovered novel prodrug that releases a potent, irreversible pan-ERBB (EGFR, HER2 and HER4) TKI. It is designed to be inactive under normal oxygen conditions but undergoes fragmentations under low oxygen conditions (hypoxia) to release the potent irreversible active metabolite (tarloxotinib-E) that has activity against both normal and mutant versions of the ERBB family. Selective production of tarloxotinib-E under hypoxic conditions generates a therapeutic window where it is selectively activated in hypoxic tumor regions to deliver higher drug delivery to tumor tissue. This reduces systemic exposure which avoids on-target EGFR related toxicities than standard EGFR TKI. In a mouse xenograft model of a human derived EGFR exon 20 insertion, intra-tumoral tarloxotinib-E levels were 20 time higher than skin and 50 times higher than plasma demonstrating selective tumor conversion. This strategy broadens the therapeutic window leading to improved efficacy, while reducing toxicity. Multiple pre-clinical studies have further demonstrated the efficacy of tarloxotinib compared to standard EGFR inhibitors.

Phase I clinical trials to determine the MTD and DLTs of tarloxotinib enrolled 27 patients with locally advanced or metastatic solid tumors. Of the patients that received tarloxotinib as a weekly 1-hour infusion, 6 patients received the drug at the recommended Phase 2 dose of 150 mg/m2 with good tolerance.

The combination of tarloxotinib with sotorasib is poised to provide highly specific tumor inhibition while targeting the vertical KRAS signaling pathway with minimal toxicity. The combination is unlikely to result in clinically relevant drug-drug interaction (DDI) based on absorption, metabolism, elimination or protein-binding. Tarloxotinib is intravenously administered while sotorasib is a small molecule that is administered orally; no absorption interactions are expected.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of squamous or non-squamous NSCLC with KRAS G12C mutation
2. Unresectable or metastatic disease
3. No available treatment with curative intent
4. Must have previously received treatment with at least a platinum-containing chemotherapy regimen
5. Must have previously received at least one month trial of sotorasib or a therapy targeting KRAS G12C mutation with documented progression. If sotorasib dose from prior therapy was reduced for toxicity, patients that meet the above criteria are expected to receive study treatment at the reduced dose.
6. Must have measurable or evaluable disease as defined by RECIST 1.1
7. Age >18 years
8. Life expectancy of at least 3 months
9. Recovery from adverse effect of prior therapy at the time of enrollment
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
11. Laboratory values within the screening period:

    1. Absolute neutrophile count > 1000/mm3
    2. Platelet count > 100,000 /mm3
    3. Hemoglobin > 8 in the absence of transfusions for at least 2 weeks
    4. Total bilirubin < 1.5 x upper limit of normal (or < 3 x ULN if associated with liver metastases or Gilbert's disease)
    5. Aspartate transaminase (AST) or alanine transaminase (ALT) < 3 x ULN (or < 5x ULN if associated with liver metastases
    6. Creatinine clearance (CrCl) > 60 mL/min
12. Women of child-bearing potential agrees to use contraception while participating in the study and for a period of 6 months following termination of study treatment
13. Completed informed consent process
14. Willing to comply with clinical trial instructions and requirements.

Exclusion Criteria:

1. Active brain metastases. Patients are eligible if brain metastases are asymptomatic measuring no more than 2.0 cm each and confined to the cerebral hemispheres if neurologically stable and must be on a stable or tapering dose of corticosteroids for at least 2 weeks prior to C1D1.
2. History of intestinal disease or major gastric surgery likely to alter absorption of study treatment or inability to swallow pills
3. Congestive heart failure > NYHA Class 3
4. QTc > 480 milliseconds or family history of Long QT syndrome
5. Ongoing need for a medication with a known risk of Torsades de Pointes that cannot be switched to alternative treatment prior to study entry.
6. Pregnancy or breast feeding
7. Has known activating oncogene-driver mutations, including but not limited to KRAS, ALK, ROS1, RET, BRAF, NTRK1/2/3, MET, EGFR
8. Previously have received anti-EGFR or anti-HER2 TKIs
9. Previously have received anti-EGFR or anti-HER2 monoclonal antibodies
10. Clinically active or symptomatic interstitial lung disease
11. AST and ALT>3xULN if no hepatic metastases are present; >5xULN if hepatic metastases are present; total bilirubin >1.5xULN; 3xULN with direct bilirubin >1.5 x ULN in the presence of Gilbert's syndrome
12. Known concurrently malignancy that is expected to require active treatment within 2 years or may interfere with the interpretation of the efficacy and safety outcomes of this study.
13. Infection requiring systemic treatment within 7 days prior to cycle 1 day1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants in Stage 1 received the same dose of Tarloxotinib (150 mg/m² weekly) following initial safety evaluation. Therefore, participants were combined into a single arm/group in the Participant Flow table to reflect this uniform dosing. All 5 patients were enrolled only into the starting dose, Dose Level 0 (full dose: 960 mg Sot; 150 mg/m2 Tarlox).
Groups:
- STAGE 1: SAFETY LEAD IN (n=6-18, depending on number of DLs explored): SAFETY LEAD IN (n=6-18, depending on number of DLs explored) 3+3 design dependent on DLTs - Participants receive the same dose at start of safety lead-in and if too much toxicity, then the participant steps down to the next lowest dose.
  Sotorasib and Tarloxotinib: Sotorasib 960 mg PO daily + tarloxotinib 150 mg/m2 IV weekly
  Sotorasib and Tarloxotinib: Sotorasib 960 mg PO daily + tarloxotinib IV weekly at the combination RP2D (RP2Dc).
Period: Overall Study
Arm/Group | STAGE 1: SAFETY LEAD IN (n=6-18, depending on number of DLs explored) | STAGE 2: EFFICACY (n=12)
Started | 5 | 0
Completed | 4 | 0
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Study was prematurely terminated due to study drug being withdrawn by manufacturer.
Groups:
- Total: Total of all reporting groups
Arm/Group | STAGE 1: SAFETY LEAD IN (n=6-18, Depending on Number of DLs Explored) | STAGE 2: EFFICACY (n=12) | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Continuous [Mean (Full Range); unit: years] | 59 [51 to 85] |  | 59 [51 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 5 |  | 5
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 4 |  | 4
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Objective Response
Description: (OR = CR+PR) measured by CT and assessed per RECIST 1.1. Complete response (CR) and partial response (PR) require confirmatory CT
Time Frame: There is no defined time frame for response assessment in the protocol. Presumably, patients are followed for response until the they stop taking study drug and/or have disease progression. The latest an assessment occurred for a patient was 40 weeks.
Population: Subjects only enrolled in safety-lead in there is no data for efficacy portion. Study was prematurely terminated due to study drug being withdrawn by manufacturer. No patient had an Objective Response to therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | STAGE 1: SAFETY LEAD IN (n=6-18, depending on number of DLs explored) | STAGE 2: EFFICACY (n=12)
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

2. Secondary Outcome: Duration of Response
Description: measured from the date of first response (CR or PR) to date of disease progression (taking as reference for progressive disease the smallest measurements recorded since the treatment started) or death.
Time Frame: At least 4 weeks.
Population: Study was prematurely terminated due to study drug being withdrawn by manufacturer. Patients can have a response at one time point but at the next time point data was not collected to confirm which is necessary to measure duration of response.
Measure: Count of Participants; unit: Participants
Arm/Group | STAGE 1: SAFETY LEAD IN (n=6-18, depending on number of DLs explored) | STAGE 2: EFFICACY (n=12)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Disease Control Rate
Description: (DCR) based on patient who had CR or PR or Stable disease (SD)
Time Frame: Through study completion, an average of 18 months.
Population: Study was prematurely terminated due to study drug being withdrawn by manufacturer. Patients can have a response at one time point but at the next time point it was not confirmed which is necessary to measure disease control rate.
Measure: Count of Participants; unit: Participants
Arm/Group | STAGE 1: SAFETY LEAD IN (n=6-18, depending on number of DLs explored) | STAGE 2: EFFICACY (n=12)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Best Overall Response
Description: (BOR) determined from a sequence of responses assessed. Two objective status determinations of CR before progression are required for a BOR of CR. Two determinations of PR or better before progression, but not qualifying for a CR, are required for a BOR of PR.
Time Frame: A minimum timeframe of 8 weeks is required for a BOR of SD.
Population: No participants could be observed for BOR. Study was prematurely terminated due to study drug being withdrawn by manufacturer.
Measure: Count of Participants; unit: Participants
Arm/Group | STAGE 1: SAFETY LEAD IN (n=6-18, depending on number of DLs explored) | STAGE 2: EFFICACY (n=12)
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

5. Secondary Outcome: Progression Free Survival
Description: (PFS) as measured from the date of first study drug dose to the date of the first objective documentation of radiographic disease progression or death due to any cause.
Time Frame: From the date of first study drug dose to the date of the first objective documentation of radiographic disease progression or death due to any cause, up to approximately 100 months.
Population: There were no number of events obtained to be observed for PFS. Study was prematurely terminated due to study drug being withdrawn by manufacturer.
Measure: Count of Participants; unit: Participants
Arm/Group | STAGE 1: SAFETY LEAD IN (n=6-18, depending on number of DLs explored) | STAGE 2: EFFICACY (n=12)
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

6. Secondary Outcome: Overall Survival
Description: (OS) as measured from the date of first study drug dose to the date of death by any cause.
Time Frame: Follow-up for survival continues until 6 months after the last patient on-study visit.
Population: One participant was not evaluable due to death before receiving first dose of study drug. Study was terminated early due to study drug being withdrawn by manufacturer.
Measure: Median (Full Range); unit: years
Arm/Group | STAGE 1: SAFETY LEAD IN (n=6-18, depending on number of DLs explored) | STAGE 2: EFFICACY (n=12)
Number analyzed (Participants) | 4 | 0
years | 0.75 [0.00 to 0.75] |

ADVERSE EVENTS:
Time Frame: Up to 22 months
Description: No participants were enrolled in Stage 2 of the study. Study was prematurely withdrawn due to study drug being withdrawn by manufacturer.
Arm/Group | STAGE 1: SAFETY LEAD IN (n=6-18, depending on number of DLs explored) | STAGE 2: EFFICACY (n=12)
All-Cause Mortality (participants affected / at risk) | 1/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/0
Other Adverse Events (participants affected / at risk) | 4/4 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STAGE 1: SAFETY LEAD IN (n=6-18, depending on number of DLs explored) (N=4) | STAGE 2: EFFICACY (n=12) (N=0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Nausea (Gastrointestinal disorders) | 1 (1) | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STAGE 1: SAFETY LEAD IN (n=6-18, depending on number of DLs explored) (N=4) | STAGE 2: EFFICACY (n=12) (N=0)
Prolonged QTc interval (Cardiac disorders) | 2 (2) | NA
Anorexia (Metabolism and nutrition disorders) | 2 (2) | NA
Dizziness (Nervous system disorders) | 2 (2) | NA
Fatigue (General disorders) | 2 (2) | NA
Hypotension (Vascular disorders) | 2 (2) | NA
Diarrhea (Gastrointestinal disorders) | 2 (2) | NA
Facial muscle weakness (Nervous system disorders) | 1 (1) | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA
Otitis media (Infections and infestations) | 1 (1) | NA
Allergic reaction (Immune system disorders) | 1 (1) | NA
Gait disturbance (General disorders) | 1 (1) | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | NA
Cardiac chest pain (Cardiac disorders) | 1 (1) | NA
Dysuria (Renal and urinary disorders) | 1 (1) | NA
Hematuria (Renal and urinary disorders) | 1 (1) | NA
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | NA
Constipation (Gastrointestinal disorders) | 1 (1) | NA
Gastroesophageal reflux disease (GERD) (Gastrointestinal disorders) | 1 (1) | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | NA
Limb edema (Skin and subcutaneous tissue disorders) | 1 (1) | NA
Umbilical hernia (Skin and subcutaneous tissue disorders) | 1 (1) | NA

LIMITATIONS AND CAVEATS:
1 participant died prior to first dose of study drug due to existing comorbidity complications and was non-evaluable. Study was prematurely terminated due to study drug being withdrawn by manufacturer. Overall survival calculation influenced by one participant that withdrew consent for follow-up at the time of end of study treatment and admission to hospice care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT05313009/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT05313009/ICF_001.pdf